CLINICAL TRIAL: NCT04144504
Title: Prospective Randomized Controlled Trial on Balloon Dilatation and Plastic Stenting Versus Retrievable Metallic Stenting for Biliary Anastomotic Stricture After Liver Transplantation
Brief Title: Plastic Stenting Versus Retrievable Metallic Stenting for Biliary Anastomotic Stricture After Liver Transplantation
Acronym: LT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Siu-Ho Chok, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 19-006
Record Dates: First submitted 2019-10-09; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Biliary Anastomotic Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plastic stenting (Active Comparator): Patients with post-liver transplantation and suffer from biliary anastomotic stricture would be given balloon dilatation and plastic stenting for treatment.
  Interventions: Device: Plastic stenting
- Retrievable metallic stenting (Active Comparator): Patients with post-liver transplantation and suffer from biliary anastomotic stricture would be given retrievable metallic stenting for treatment.
  Interventions: Device: Retrievable metallic stenting

INTERVENTIONS:
Device: Retrievable metallic stenting — Use of retrievable metallic stents for the treatment of biliary anastomotic stricture after liver transplantation
  Arms: Retrievable metallic stenting
Device: Plastic stenting — Use of plastic stents
  Arms: Plastic stenting

SUMMARY:
Liver transplantation is the best treatment option for patients with end-stage liver disease and early unresectable hepatocellular carcinoma. Unfortunately, biliary complication after liver transplantation is still the Achilles' heel, especially in living donor liver transplantation. Early treatment with endoscopy can achieve satisfactory outcomes. Most of the time, biliary anastomotic stricture can be treated by endoscopic retrograde cholangiopancreatography with balloon dilatation with or without plastic stent insertion. Although endoscopic treatment has been reported to have a successful rate of over 70%, multiple sessions of endoscopic treatment, typically 4 to 5 sessions, are frequently required before adequate stricture dilatation is achieved. This is likely secondary to suboptimal post-dilatation splintage. The most common and popular form of splintage is plastic stent insertion. Unfortunately, plastic biliary stent has a small calibre, and therefore even with multiple stents the configuration of buttressing would not provide a circumferential, evenly distributed buttressing effect at the dilated stricture site. Moreover, given the small calibre of the plastic stent, there is higher resistance on the inner surface of the stent, leading to a higher chance of stent blockage. Many studies have suggested that self-expandable metallic stent (SEMS) is superior to plastic stent in terms of patency rate. However, SEMS is generally reserved for malignant stricture due to its permanent nature, as the traditional SEMS is not removable. Recently, retrievable SEMS (r-SEMS) has been developed, and its indications have been extended to include benign disease conditions. It has been reported that a series of 29 patients with biliary anastomotic stricture treated by r-SEMS, and they concluded that r-SEMS was safe and efficacious. Results of the preliminary study on 5 patients at our centre were favourable; all of the patients had no stricture after retrievable metallic stenting for at least 3 months and no complication was encountered.

DETAILED DESCRIPTION:
Biliary anastomotic stricture (BAS) is one of the most common complications after liver transplantation (LT). It happens more often after living donor liver transplantation (LDLT) than deceased donor liver transplantation (DDLT). The reported incidence was 20% in LDLT and 12% in DDLT. Although BAS seldom affects graft survival, it is associated with significant morbidity and affects quality of life. Clinical manifestation of BAS can be highly variable, ranging from low-grade cholangitis with slightly deranged liver function to life-threatening septic shock to graft and multi-organ failure. Up to 30% of the cases of BAS require surgical intervention at some point. Revision hepaticojejunostomy - a major undertaking judging from the magnitude of the operation - is sometimes required as a remedial procedure. Most of the time BAS can be treated by endoscopic retrograde cholangiopancreatography (ERCP) with balloon dilatation with or without plastic stent insertion. Although endoscopic treatment has been reported to have a successful rate of over 70%, multiple sessions of endoscopic treatment, typically 4 to 5 sessions, are frequently required before adequate stricture dilatation is achieved. This is likely secondary to suboptimal post-dilatation splintage. Since stricturoplasty features breaking up the fibrous ring at the anastomotic site and hence widening the calibre of the lumen, any new wound created by dilatation injury is susceptible to the formation of new scar. Therefore, some form of buttressing device is needed to keep the anastomotic site open. This underscores the importance of post-dilatation splintage. The most common and popular form of splintage is plastic stent insertion. Unfortunately, plastic biliary stents have a small calibre, with the largest size being Fr11.5 only. Even if multiple stents are inserted, the configuration of buttressing would not provide a circumferential, evenly distributed buttressing effect at the dilated stricture site. Moreover, given the small calibre of the plastic stent, there is higher resistance on the inner surface of the stent, leading to a higher chance of stent blockage. Frequent admissions for repeated dilatation and stent exchange (not to mention emergency admission for a cholangitic episode secondary to stent blockage) significantly disrupt the patient's normal daily activities and form a clinical and financial burden to the community. Many studies have suggested that self-expandable metallic stent (SEMS) is superior to plastic stent in terms of patency rate. However, SEMS is generally reserved for malignant stricture due to its permanent nature, as the traditional SEMS is not removable. Recently, retrievable SEMS (r-SEMS) has been developed, and its indications have been extended to include benign disease condition. It has been reported that a series of 29 BAS patients treated by r-SEMS, and they concluded that r-SEMS was safe and efficacious. Results of the preliminary study on 5 patients at our centre were favourable; all of them had no stricture for at least 4 months after r-SEMS treatment and no complication was encountered. The median number of session for success was 2, which is significantly fewer than that in the ordinary approach (median session: 4).

Up till this moment, there is no randomized controlled trial comparing the performance of r-SEMS with that of the conventional approach. In this study, the null hypothesis is that there is no difference in performance between r-SEMS and the conventional approach in endoscopic treatment of BAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give informed consent

Exclusion Criteria:

* Patients who refuse to give consent
* Patients who have previously hepaticojejunostomy as biliary re-construction
* Patients who have previous upper gastrointestinal surgery making endoscopic treatment not posssible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of endoscopic sessions to achieve resolution of stricture | Two months
  To compare the total number of treatments to successfully resolve the problem of biliary stricture in each arm
Percentage of successful treatment | Two months
  To compare the total rate of successful treatment in each arm
Pain score after treatment | Two months
  To compare the differential pain score experienced by patients in each arm as rated by facial pain score scale (Ranging from 0-10) Maximum pain score = 10; No pain = 0)
Patient's quality of life | Two months
  To compare the quality of life as experienced by patients who have undergone stenting treatment(s) in each arm using SF36 questionnaire with maximum score=100 as the best outcome and minimum score=0 as the worst

SECONDARY OUTCOMES:
Complication rate | 2 months
  To compare the rate of complications such as post-ERCP pancreatitis, bleeding and perforation between patients who have received plastic or metallic stents
Hospital stay | Two months
  To compare the duration of hospital stay between patients who have received plastic or metallic stents
BAS recurrence | Two months
  To compare the rate of BAS recurrence between patients who have received plastic or metallic stents
Readmission rate | Two months
  To compare the rate of readmission rate between patients who have received plastic or metallic stents

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chok, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Akamatsu N, Sugawara Y, Hashimoto D. Biliary reconstruction, its complications and management of biliary complications after adult liver transplantation: a systematic review of the incidence, risk factors and outcome. Transpl Int. 2011 Apr;24(4):379-92. doi: 10.1111/j.1432-2277.2010.01202.x. Epub 2010 Dec 10. PMID 21143651
- [Background] Sundaram V, Jones DT, Shah NH, de Vera ME, Fontes P, Marsh JW, Humar A, Ahmad J. Posttransplant biliary complications in the pre- and post-model for end-stage liver disease era. Liver Transpl. 2011 Apr;17(4):428-35. doi: 10.1002/lt.22251. PMID 21445926
- [Background] Castaldo ET, Pinson CW, Feurer ID, Wright JK, Gorden DL, Kelly BS, Chari RS. Continuous versus interrupted suture for end-to-end biliary anastomosis during liver transplantation gives equal results. Liver Transpl. 2007 Feb;13(2):234-8. doi: 10.1002/lt.20986. PMID 17256781
- [Background] Johnson MW, Thompson P, Meehan A, Odell P, Salm MJ, Gerber DA, Zacks SL, Fried MW, Shrestha R, Fair JH. Internal biliary stenting in orthotopic liver transplantation. Liver Transpl. 2000 May;6(3):356-61. doi: 10.1053/lv.2000.5303. PMID 10827239
- [Background] Mahajani RV, Cotler SJ, Uzer MF. Efficacy of endoscopic management of anastomotic biliary strictures after hepatic transplantation. Endoscopy. 2000 Dec;32(12):943-9. doi: 10.1055/s-2000-9619. PMID 11147942
- [Background] Buxbaum JL, Biggins SW, Bagatelos KC, Ostroff JW. Predictors of endoscopic treatment outcomes in the management of biliary problems after liver transplantation at a high-volume academic center. Gastrointest Endosc. 2011 Jan;73(1):37-44. doi: 10.1016/j.gie.2010.09.007. Epub 2010 Nov 12. PMID 21074761
- [Background] Tabibian JH, Asham EH, Han S, Saab S, Tong MJ, Goldstein L, Busuttil RW, Durazo FA. Endoscopic treatment of postorthotopic liver transplantation anastomotic biliary strictures with maximal stent therapy (with video). Gastrointest Endosc. 2010 Mar;71(3):505-12. doi: 10.1016/j.gie.2009.10.023. PMID 20189508
- [Background] Graziadei IW, Schwaighofer H, Koch R, Nachbaur K, Koenigsrainer A, Margreiter R, Vogel W. Long-term outcome of endoscopic treatment of biliary strictures after liver transplantation. Liver Transpl. 2006 May;12(5):718-25. doi: 10.1002/lt.20644. PMID 16482553
- [Background] Pasha SF, Harrison ME, Das A, Nguyen CC, Vargas HE, Balan V, Byrne TJ, Douglas DD, Mulligan DC. Endoscopic treatment of anastomotic biliary strictures after deceased donor liver transplantation: outcomes after maximal stent therapy. Gastrointest Endosc. 2007 Jul;66(1):44-51. doi: 10.1016/j.gie.2007.02.017. PMID 17591473
- [Background] Morelli J, Mulcahy HE, Willner IR, Cunningham JT, Draganov P. Long-term outcomes for patients with post-liver transplant anastomotic biliary strictures treated by endoscopic stent placement. Gastrointest Endosc. 2003 Sep;58(3):374-9. doi: 10.1067/s0016-5107(03)00011-7. PMID 14528211
- [Background] Deviere J, Nageshwar Reddy D, Puspok A, Ponchon T, Bruno MJ, Bourke MJ, Neuhaus H, Roy A, Gonzalez-Huix Llado F, Barkun AN, Kortan PP, Navarrete C, Peetermans J, Blero D, Lakhtakia S, Dolak W, Lepilliez V, Poley JW, Tringali A, Costamagna G; Benign Biliary Stenoses Working Group. Successful management of benign biliary strictures with fully covered self-expanding metal stents. Gastroenterology. 2014 Aug;147(2):385-95; quiz e15. doi: 10.1053/j.gastro.2014.04.043. Epub 2014 May 4. PMID 24801350
- [Background] Chok KS, Chan SC, Cheung TT, Sharr WW, Chan AC, Fan ST, Lo CM. A retrospective study on risk factors associated with failed endoscopic treatment of biliary anastomotic stricture after right-lobe living donor liver transplantation with duct-to-duct anastomosis. Ann Surg. 2014 Apr;259(4):767-72. doi: 10.1097/SLA.0b013e318294d0ce. PMID 23657086
- [Background] Tee HP, James MW, Kaffes AJ. Placement of removable metal biliary stent in post-orthotopic liver transplantation anastomotic stricture. World J Gastroenterol. 2010 Jul 28;16(28):3597-600. doi: 10.3748/wjg.v16.i28.3597. PMID 20653071